CLINICAL TRIAL: NCT04786483
Title: The Effect of Laughter Therapy on Students' Anxiety, Life Satisfaction and Psychological Well-being in the Covid-19 Pandemic
Brief Title: The Effect of Laughter Therapy on Students in the COVID-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: Prof. Dr. Şule Ecevit Alpar (Unknown)
Responsible Party: Principal Investigator, Canan Eraydın, Lecturer, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021/06
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Laughter Yoga; Anxiety; Life Satisfaction; Psychological Well-being; COVID-19
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction; Psychological Well-Being; COVID-19 | interventions — Mutation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Therapy group (Experimental): All students enrolled in the laughter therapy group will receive a total of 10 sessions of laughter therapy, 60 minutes, 2 days a week.
  Interventions: Other: Laughter Theraphy
- Control (No Intervention): No attempt will be made to students in this group.

INTERVENTIONS:
Other: Laughter Theraphy — Laughter therapy will be applied for 60 minutes, 10 sessions, 2 days a week. The therapy, which starts with the stimulation of the acupuncture points in the palm and acquaintance with hand clapping for an average of 10 minutes, continues with deep breathing and breathing exercises that include diaphragmatic breathing. The childish games section, which is played to reveal and trigger simulated laughter, is the section where laughter starts as "if" and turns into reality. The last part is the part where the group makes eye contact for no reason and for no reason, and laughs for at least 3 minutes unconditionally. In the last part, wish meditation and relaxation sessions are performed.
  Other Names: Alternative
  Arms: Laughter Therapy group

SUMMARY:
This study was designed as a randomized controlled, pre-test-post-test control group in order to determine the effect of laughter therapy on anxiety, life satisfaction and psychological well-being of nursing students. Laughter therapy was applied to the experimental group for at least 60 minutes, 10 sessions two days a week. For the evaluation, the state-continuity anxiety scale, life satisfaction scale, psychological well-being scale were applied at the pre-application stage (pre-test) and after the laughter therapy sessions (post-test). The following hypotheses were included in this study;

H1: Laughter therapy given during the Covid19 pandemic reduces the anxiety level of intern students.

H2: Laughter therapy given during the Covid19 pandemic affects the life satisfaction of intern students.

H3: During the Covid19 pandemic process, the laughter therapy given to interns affects the relationship between anxiety levels and life satisfaction.

H4: Laughter therapy given to intern students during the Covid19 pandemic process affects psychological well-being.

DETAILED DESCRIPTION:
Today, all countries are struggling with COVID-19, which typically presents with mild symptoms but causes serious mortality in the world population. In addition to the routine changes due to the pandemic, face-to-face education has been switched to online education. The integration of online education and more technology into the curriculum than ever before has increased students' anxiety towards learning. It was also found to cause high levels of anxiety and stress, characterized by feelings of risk, insecurity, and unhappiness. Studies show that high levels of anxiety negatively affect students' adaptation to daily life and their life satisfaction levels. In recent years, non-pharmacological techniques have been widely used in reducing anxiety and stress. One of them is laughter therapy. Laughter therapy reduces feelings of negative stress, anxiety, and depression by increasing the body's readiness to deal with different types of problems. The aim of this study is to examine the effects of online laughter therapy on anxiety, life satisfaction and psychological well-being levels of nursing students, who have switched to online education during the pandemic process.

ELIGIBILITY:
Inclusion Criteria:

* A student of the Faculty of Health Sciences, Department of Nursing and enrolled in the fall semester,
* Who has not studied laughter yoga before or did not do laughter yoga,
* It will create students who agree to participate in the research.

Exclusion Criteria:

* Being a foreign national,
* Having a situation where laughter yoga is not recommended (having surgery in the abdominal region in the last three months, uncontrolled hypertension, chronic cough, incontinence, acute back pain, acute mental disorders, consumption of antipsychotic drugs, glaucoma, hernia, epilepsy),
* Students with simultaneous participation in any complementary treatment methods will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-10 (Estimated)

PRIMARY OUTCOMES:
psychological well-being | 4 months
  What are the anxiety levels of the students after the laughter therapy given during the Covid19 pandemic? State and trait anxiety scales will be used to measure students' anxiety levels before and after laughter therapy. The scale is a Likert-type scale that separately measures state-continuity anxiety levels with 20 questions. The scale consists of twenty-item state anxiety and trait anxiety scales, with high scores showing high levels of anxiety, and low scores showing low levels of anxiety. The total score obtained from both scales varies between 20-80. Big score indicates high anxiety level, small score indicates low anxiety level. It is a four-degree scale ranging from "None" to "Totally".
life satisfaction | 4 months
  What is the life satisfaction of the students after the laughter therapy given during the Covid19 pandemic? The life satisfaction levels of the students before and after the laughter therapy will be measured using the 'life satisfaction scale'.
  The scale consists of five positive statements. The scale, which aims to measure general life satisfaction, is suitable for all ages, from adolescents to adults. The scale has a 7-point Likert type evaluation. Level of participation in scale items "1 = Not at all appropriate", "2 = Not suitable", "3 = Somewhat unsuitable", "4 = Neither suitable nor not appropriate", "5 = Somewhat appropriate", "6 = Not suitable", It is scored as "7 = Very suitable". A minimum of 5 and a maximum of 35 points can be obtained from scale items. A low score on the scale is accepted as an indicator of low life satisfaction.
Psychological Well-being | 4 months
  What are the psychological well-being levels of the students after the laughter therapy given during the Covid19 pandemic? Psychological well-being scale will be used to evaluate students' psychological well-being before and after laughter therapy.
  Psychological well-being scale consists of eight items. The scale is scored between 1-7. The high score to be obtained from the scale indicates that the person has psychological power.

CONTACTS AND LOCATIONS:
Overall Officials: Şule Ecevit Alpar, Doctorate, Study Director — Üniversite
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morishima T, Miyashiro I, Inoue N, Kitasaka M, Akazawa T, Higeno A, Idota A, Sato A, Ohira T, Sakon M, Matsuura N. Effects of laughter therapy on quality of life in patients with cancer: An open-label, randomized controlled trial. PLoS One. 2019 Jun 27;14(6):e0219065. doi: 10.1371/journal.pone.0219065. eCollection 2019. PMID 31247017
- [Background] Kuru Alici N, Zorba Bahceli P, Emiroglu ON. The preliminary effects of laughter therapy on loneliness and death anxiety among older adults living in nursing homes: A nonrandomised pilot study. Int J Older People Nurs. 2018 Dec;13(4):e12206. doi: 10.1111/opn.12206. Epub 2018 Jul 13. PMID 30004172
- [Result] Sahu P. Closure of Universities Due to Coronavirus Disease 2019 (COVID-19): Impact on Education and Mental Health of Students and Academic Staff. Cureus. 2020 Apr 4;12(4):e7541. doi: 10.7759/cureus.7541. PMID 32377489